CLINICAL TRIAL: NCT06267079
Title: Effect of Core Stability Exercise on Symmetrical Weight Bearing in Chronic Stroke Patient
Brief Title: Core Stability, Symmetrical Weight-bearing Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Arafa Abdel Halim, clinical researcher Submitted in partial fulfillment of the requirements of Master Degree in Department of Physical Therapy for Neurology Faculty of Physical Therapy Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: core stability
Record Dates: First submitted 2024-02-06; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Other): Core stability Exercises. Each participant in the group (A) underwent eighteen sessions of core stability exercises very other day for one and half months, 3 sessions /week, each session for 1hour (30 minutes for core exercises then 30 minutes Selected physical therapy program).
  + Selected physical therapy program.
  Interventions: Other: core stability exercise
- control group (Other): Selected physical therapy program. all participants in both groups (A & B) had three sessions per week for a month and a half, every other day. of Selected physical therapy program which consist of (Exercises for tone modulation, balance, lower limb muscular strengthening, and stretching)
  Interventions: Other: core stability exercise

INTERVENTIONS:
Other: core stability exercise — Each participant in the group (A) underwent eighteen sessions of core stability exercises very other day for one and half months, 3 sessions /week, each session for 1hour (30 minutes for core exercises then 30 minutes Selected physical therapy program).

SUMMARY:
To evaluate the effect of core stability exercise on symmetrical weight bearing in chronic stroke patients?

DETAILED DESCRIPTION:
Stroke is a syndrome characterized by quickly emerging clinical indicators of a focal (or global) disruption of brain function. The symptoms can last for more than 24 hours or even result in death, and there is no known reason for them other than vascular origin. Over 80% of all strokes are caused by an ischemic stroke. A large artery blockage typically results in tissue infarction, which is the non-selective loss of all brain cells in the affected areas of the brain if it is not quickly reversed. Determining the location and size of these infarcts is crucial. the long-term functional deficits resulting from ischemic stroke. After a stroke, patients' ability to bear weight symmetrically is similarly compromised; they may bear between 61 and 80% of their body weight on a non-paretic leg. Physiotherapy procedures targeted at enhancing core stability can enhance the lumbopelvic-hip musculature's strength, coordination, and endurance, potentially reducing physical deficits linked to compromised trunk function. Because these muscles are crucial for both stability and lumbar posture control (by the employment of Core stability is commonly utilized in whole-body exercises to enhance the strength of the muscles around the stomach, lumbar, and pelvic regions, whether they be tonic or postural muscles. The trunk is the body's center pivot point, serving as a vital component for functional activity, balance, postural control, and extremity coordination. Consequently, the trunk is very important. in the recovery procedure. There is a substantial body of research demonstrating that Trunk control, balance when sitting and standing, and mobility can all be improved with trunk training. in stroke patients, according to recent studies in systemic reviews. So, the purpose of the current study was to detect the effect of core stability exercise on symmetrical weight bearing in patients with chronic stroke

ELIGIBILITY:
Inclusion Criteria:

1. Forty hemiparetic patients were diagnosed and referred to by a neurologist.
2. All patients must be ambulant
3. The spasticity of lower limbs ranges from (grade 1: 1+) according to Modified Ashworth Scale.
4. Patients with sufficient cognitive abilities that enables them to understand and follow instructions (Mini-Mental Scale >24). (
5. Age ranges from 50 to 65 years in both sexes.
6. Duration of stroke was more than 6 months up to 24 months. -

Exclusion Criteria:

* The patients were excluded if they had any of the following:

  1. Musculoskeletal disorders such as severe arthritis grade (3-4) of osteoarthritis, lower limb fractures less than 6 months or contractures of fixed deformity.
  2. Cognitive impairment (a score less than 24 according to the MMSE)
  3. Patients with diabetic neuropathy.
  4. Recurrent stroke.
  5. Rheumatologic or endocrinologic disorders that may cause ROM restriction.
  6. Patients suffering from cognitive, or emotional disturbance.

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-09-05 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Each patient was assessed by Balance Berg scales pretreatment. and repeated Measurements were taken after treatment. Each patient was assessed by Digital weight scale and Balance Berg scales | six weeks
  The Berg Balance Scale (BBS) was used to assess static and dynamic balance
Each patient was assessed by Digital weight scale pre treatment and repeated Measurements were taken after treatment. | 6 week
  Digital weight scale:

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of physical therapy Cairo university, Cairo, Egypt